CLINICAL TRIAL: NCT02061150
Title: Neonatal Sepsis Workup for High Risk Newborns - Evaluation of Need and Ways to Prevent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-104-13
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Neonatal Sepsis
Keywords: Early onset GBS sepsis; Prevention; Maternal risk factors
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asymptomatic newborns that had sepsis workup: Evaluation of medical records of asymptomatic newborns that had sepsis workup in the first 48 hours of life.

SUMMARY:
Sepsis is a significant cause of morbidity and mortality among newborns. Due to strict criteria and in order to diagnose and prevent early-onset group B streptococcal (EOGBS) sepsis, many infants undergo a sepsis workup due to risk factors alone, even though they are asymptomatic. Our goal is to evaluate the number of newborns that undergo sepsis workup due to risk factors alone, to determine the number of newborns having positive blood cultures, and to establish ways to reduce the number of asymptomatic infants undergoing sepsis workup.

ELIGIBILITY:
Inclusion Criteria:

Term newborns with blood cultures taken from them the first 48 hrs

Exclusion Criteria:

* Preterm newborns
* Septic/ill appearing newborns
* Newborns requiring admission to NICU

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asymptomatic term/near term newborns to a mother with infectious risk factors such as premature rupture of membranes, GBS-carrier etc, that underwent sepsis work up due to their maternal risk factors,
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic newborns that underwent sepsis workup | 3 years
  The number of. asymptomatic newborns that underwent sepsis workup due to maternal risk factors only will be determined

SECONDARY OUTCOMES:
Positive blood cultures out of total cultures | 3 years
  Percentage of positive blood cultures out of the total cultures that were taken.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hillel Yaffe Medical Center, Hadera, Israel